CLINICAL TRIAL: NCT06726876
Title: Therapeutic Effect of Manuka Honey Oral Rinse in Periodontitis Patients Undergoing Hemodialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: R626
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis; Hemodialysis
Keywords: Manuka honey; fibroblast growth factor-21; periodontitis; hemodialysis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Treatment: Normal saline rinse.
  Protocol:
  Follow the same protocol as the intervention group but using normal saline rinses instead of Manuka honey.
  Additional Treatment: Patients will receive scaling and root debridement and locally delivered 0.5 ml non-diluted Thyme honey on sites with PPD ≥ 5 mm.
  Supplementary Care: Motivation, oral hygiene instructions (proper tooth brushing technique, flossing, interdental brush, mouthwash usage), scaling, polishing, and root debridement with an ultrasonic scaler and Gracey curettes.
  Interventions: Drug: Normal saline rinses.
- Intervention Group (Experimental): Treatment: Manuka honey oral rinse.
  Protocol:
  Applied as an oral rinse based on the Biswal et al. administration protocol.
  Patients will have oral rinses (20 ml of Manuka honey diluted in 100 ml of purified water) 3 times per day.
  Patients will be instructed not to swallow the Manuka honey oral rinse.
  Additional Treatment: Patients will receive scaling and root debridement and locally delivered 0.5 ml non-diluted Thyme honey on sites with PPD ≥ 5 mm.
  Supplementary Care: Motivation, oral hygiene instructions (proper tooth brushing technique, flossing, interdental brush, mouthwash usage), scaling, polishing, and root debridement with an ultrasonic scaler and Gracey curettes.
  Interventions: Dietary Supplement: Manuka honey oral rinse.

INTERVENTIONS:
Dietary Supplement: Manuka honey oral rinse. — Name: Manuka Honey Oral Rinse
  Description:
  Dosage: Patients will use 20 ml of Manuka honey diluted in 100 ml of purified water.
  Administration: Oral rinse, performed 3 times per day.
  Instructions: Patients are instructed to rinse their mouths with the solution for a specified duration and avoid swallowing it.
  Unique Elements:
  Active Ingredient: Manuka honey, known for its unique antibacterial properties due to high levels of methylglyoxal (MGO).
  Mechanism of Action: MGO and Non-Peroxide Activity (NPA) contribute to antibacterial potency, effective against antibiotic-resistant bacteria, and potential immunomodulatory effects that aid wound healing and tissue regeneration.
  Additional Procedures: Scaling and root debridement, along with the local application of 0.5 ml non-diluted Thyme honey on sites with Probing Pocket Depth (PPD) ≥ 5 mm.
  Supplementary Care: Patients receive motivation and detailed oral hygiene instructions (proper tooth brushing technique, flossing, use of inte
  Arms: Intervention Group
Drug: Normal saline rinses. — Dosage: Patients will use 20 ml of normal saline.
  Administration: Oral rinse, performed 3 times per day.
  Instructions: Patients are instructed to rinse their mouths with the saline solution for a specified duration and avoid swallowing it.
  Unique Elements:
  Control Comparison: Provides a placebo comparison to evaluate the efficacy of the Manuka honey intervention.
  Additional Procedures: Scaling and root debridement, along with the local application of 0.5 ml non-diluted Thyme honey on sites with Probing Pocket Depth (PPD) ≥ 5 mm.
  Arms: Control Group

SUMMARY:
Chronic Kidney Disease (CKD) has a strong association with chronic periodontitis, an oral disease causing tooth loss linked to inflammation and malnutrition. While periodontitis affects 12.7% of the general population, its prevalence can rise to 39% in certain racial groups, and a dose-response relationship exists with CKD. End Stage Renal Disease (ESRD) patients show a prevalence of periodontitis ranging from 29% to 85.6%. Uremia, immunosuppression, and vitamin D deficiency are suggested factors in the etiology of periodontitis in CKD patients, with uremic toxins potentially altering the oral ecosystem.

Periodontitis involves bacterial biofilm and Gram-negative anaerobes as primary etiological factors. The main treatment goal is to reduce periodontal pathogens and control inflammation, with non-surgical periodontal therapy (NSPT) being the standard. Although various adjuncts like antibiotics and antiseptics are suggested, recent guidelines only recommend certain locally administered agents and systemic antibiotics for specific groups due to increasing bacterial resistance.

Alternative treatments like honey have gained interest, particularly Manuka honey, known for its antibacterial properties against antibiotic-resistant bacteria. This honey's effectiveness is due to its high sugar concentration, low pH, and formation of hydrogen peroxide. Manuka honey's unique component, methylglyoxal (MGO), is a potent bactericide, virucide, and fungicide, linked to its Non-Peroxide Activity (NPA) and Unique Manuka Factor (UMF) rating. MGO also has immunomodulatory effects beneficial for wound healing and tissue regeneration.

Previous studies show Manuka honey as a promising adjunct in NSPT, improving outcomes significantly without adverse effects. Ongoing research aims to evaluate its effects in ESRD patients on hemodialysis, focusing on clinical attachment levels, other periodontal parameters, and FGF 21 levels in gingival crevicular fluid.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is associated with a high prevalence of chronic periodontitis, an infectious oral disease that causes tooth loss and is linked to inflammation and malnourishment [1]. The frequency of periodontitis is 12.7% in the general population, according to recent epidemiological studies [2], but it can reach as high as 39% in certain racial groups [3, 4], and there is a dose-response relationship with CKD [5]. The prevalence of periodontitis in End Stage Renal Disease (ESRD) has been reported in smaller studies to range from 29 to 85.6% [6, 7, 8]. It has been proposed that uremia and associated immunosuppression, as well as vitamin D deficiency, play a role in the etiology of periodontitis in CKD [5, 9, 10].

Uremic toxins may potentially alter the oral ecosystem (hydrolysis of urea results in alkaline pH) promoting the growth of periodontal pathogens, in a similar manner to the demonstrated uremia-related changes in the gut environment [11, 12]. Studies using microbiological methods of limited scope have shown that ESRD individuals with periodontitis have increased levels of periodontal pathogens as compared to non-CKD controls [13].

Periodontitis is a chronic inflammatory disease affecting the teeth's supporting apparatus. Bacterial biofilm and the associated periodontal pathogenic bacteria, mainly Gram-negative anaerobes, are the main etiological factor of the disease [14].

The main goal of periodontal treatment is to reduce the number of periodontal pathogens and arrest the inflammatory process. The contemporary gold treatment standard is non-surgical periodontal therapy (NSPT), which involves scaling and root planning using manual and machine-driven (sonic or ultrasonic) instruments [15].

Various systemically administered and locally delivered adjuncts to NSPT have been suggested, including systemic and local antibiotics, antiseptics, probiotics, lasers, and photodynamic treatment. However, the latest guidelines on the treatment of periodontitis stage I-III do not support the use of adjuncts. The exception in terms of open recommendations is given for locally administered sustained-release chlorhexidine and antibiotics and the use of systemic antibiotics in specific patient groups [15].

The fact that bacteria are becoming increasingly resistant to antibiotics and antiseptics has shifted the interest of medicine to alternative treatment methods against which bacterial resistance cannot be developed. This approach includes using honey, which is increasingly used in medicine. Since the 1990s, when the first studies appeared on the therapeutic effects of honey, particular interest has been focused on its antibacterial properties against infections and antibiotic-resistant bacteria. This effect is consequential mainly of the high sugar concentration of honey, its low pH value, and the formation of hydrogen peroxide that occurs in the enzymatic breakdown of glucose by the glucose oxidase enzyme [16]. Contemporary research on the effects of honey focuses predominantly on one specific honey type, leading to the medicinal use of Manuka honey due to its antibacterial properties [17]. This is an endemic type of honey produced by bees in Australia and New Zealand from the flowers of the plant Leptospermum scoparium [18].

The concentration of hydrogen peroxide in Manuka honey is lower than in other types of honey [19]. The specific antibacterial activity in Manuka honey is based on methylglyoxal (MGO), a compound proven to be a very efficient bactericide, virucide, and fungicide. Furthermore, Manuka honey is highly effective against antibiotic-resistant bacteria [20].

The antibacterial potency of Manuka honey was found to be related to its Non-Peroxide Activity (NPA), trademarked as Unique Manuka Factor (UMF) rating, a classification system which reflects the equivalent concentration of phenol (%, w/v) required to produce the same antibacterial activity as honey, and it is correlated with the methylglyoxal and total phenols content [21]. In addition to its antimicrobial properties, published literature suggests that MGO also has immunomodulatory effects which may positively impact wound healing and tissue regeneration [22,23].

A previous pilot study indicated a promising potential of Manuka honey as an adjunct in NSPT. Despite the improvement in outcomes appearing modest in absolute terms, it was statistically significant for all follow-up time points, indicating the potential use of Manuka honey as a simple and affordable adjunct to non-surgical periodontal therapy. Furthermore, the product is considered a safe adjunct and no adverse events related to its use were reported during the study period. Encouraging results from this pilot study led to a further randomized clinical study on a larger sample that is currently being performed by our group [24].

Manuka honey oral rinse has not yet been investigated as a possible adjunct to NSPT in ESRD patients on regular hemodialysis. Therefore, this study aims to evaluate the effects of Manuka honey oral rinse on clinical attachment level (CAL) as a primary objective, and other periodontal parameters like (BOP, plaque index), and its effect on the levels of FGF 21 in gingival crevicular fluid as secondary objectives after nonsurgical periodontal treatment in patients with periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, aged above 18 years.
* All patients must be clinically diagnosed of ESRD undergoing hemodialysis.
* All patients must have a periodontal disease.
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* Smoking, Alcohol.
* Patient with history of any serious illness as malignancy, who undergo kidney transplant.
* Patients with any autoimmune disease.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) | Evaluated at baseline, 3 months, and 6 months post-treatment.
  Description: Measurement of the attachment level of the periodontal ligament to the tooth surface, indicating the health of periodontal tissues.

SECONDARY OUTCOMES:
Bleeding on Probing (BOP) | Evaluated at baseline, 3 months, and 6 months post-treatment.
  Description: Assessment of bleeding on probing, which is an indicator of inflammation in periodontal tissues.
Plaque Index | Evaluated at baseline, 3 months, and 6 months post-treatment.
  Measurement of the amount of dental plaque on the tooth surface, which is an indicator of oral hygiene.
Fibroblast Growth Factor 23 (FGF 23) Levels in Gingival Crevicular Fluid (GCF) | Evaluated at baseline and at 6 months post-treatment.
  Measurement of FGF 23 levels in gingival crevicular fluid, which may reflect tissue response and inflammation levels.
Fibroblast Growth Factor 23 (FGF 23) Levels in serum | Evaluated at baseline and at 6 months post-treatment.
  Measurement of FGF 23 levels in serum, which may reflect tissue response and inflammation levels.
Oral Health Impact Profile (OHIP-14) scores | baseline, and 6 months
  measured on a 5-point Likert scale. Lower scores indicate better oral health-related quality of life (OHRQoL)
Serum C-Reactive Protein (CRP) | baseline, 6 months
  Serum C-reactive protein (CRP) was measured as a marker of systemic inflammation in patients with end-stage renal failure (ESRF) and periodontitis. Venous blood samples were collected under standardized conditions, and serum was separated by centrifugation. CRP levels were quantified using a validated laboratory assay according to routine clinical laboratory protocols, and results were expressed in milligrams per liter (mg/L).
  CRP is an acute-phase protein produced by the liver in response to inflammatory stimuli. In ESRF, CRP levels may be chronically elevated due to uremia and dialysis-related inflammation, while periodontitis represents an additional source of persistent inflammatory burden. Accordingly, CRP in this study was used as an indicator of overall systemic inflammation rather than a disease-specific diagnostic marker. Higher CRP values were interpreted as reflecting increased inflammatory activity and were analyzed in relation to periodontal status and disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha hospital, Banhā, Egypt